CLINICAL TRIAL: NCT05142280
Title: Actively Choosing How to Cope With an Increased Risk of Cardiovascular Disease: A Randomised Web-Based Experiment
Brief Title: Active Choice Regarding Cardiovascular Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Lorraine Landais, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021.0676
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases
Keywords: Prevention; Active choice; Decision-making
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Web-based randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active choice (Experimental): This intervention contains information and an assignment to foster an active choice regarding coping with an increased CVD risk. Participants will be presented a hypothetical 'heart age' of 16 years older than their actual age. They will be asked to imagine that this heart age really applies to them. Next, participants will receive information about the meaning of the risk, including its causes and potential consequences, and about four coping strategies: changing one's lifestyle; taking medication; doing both; or changing nothing. The pros and cons of each strategy will be presented, followed by a value-clarification exercise.
  Interventions: Other: Decision-aid for cardiovascular disease risk
- Control (Other): The control group will receive online information and advice that resembles GP's usual care. The information contains a hypothetical CVD risk: a risk of 31% to get CVD within 10 years. They will be asked to imagine that this risk really applies to them. Participants will read about an imaginary GP who advices to change one's lifestyle (i.e., quitting smoking; healthy diet; more physical activity), and to use medication to decrease the risk.
  Interventions: Other: Control

INTERVENTIONS:
Other: Decision-aid for cardiovascular disease risk — The active choice intervention aims to promote an active choice regarding coping with an increased risk of cardiovascular disease. This means that individuals should (a) become aware of a discrepancy between the current and desired situation; (b) understand what the CVD risk means, and what its causes and consequences are; (c) evaluate the pros and cons of the different options to cope with the risk; and (d) are clear about their values regarding the choice.
  Other Names: Active choice intervention for cardiovascular disease risk
  Arms: Active choice
Other: Control — The control condition contains information that resembles usual care by a GP regarding CVD prevention
  Other Names: Usual Care
  Arms: Control

SUMMARY:
In this web-based RCT, the investigators will investigate whether promoting an active choice regarding coping with an increased CVD risk results in better psychological outcomes (e.g., degree of active choice; commitment toward the chosen option) compared to usual care (i.e., a GP's advice to change one's lifestyle and take medication). By 'active choice' the investigators mean a conscious and autonomous choice in which an individual (a) becomes aware of a discrepancy between the current and desired situation; (b) understands what his/her CVD risk means, and what its causes and consequences are; (c) evaluates the pros and cons of the different options to cope with the risk; and (d) is clear about his/her values regarding the choice. The different options to cope with an increased CVD risk include: changing one's lifestyle; taking medication; doing both; or changing nothing.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) continues to be a leading cause of mortality among adults. Adults at increased risk of cardiovascular disease are usually advised by their general practitioner (GP) to change their lifestyle (i.e., quit smoking; eat healthier; become more physically active). In addition, GP's regularly advice their patients to take antihypertensive and/or lipid lowering medication to decrease the CVD risk. Previous research has shown that many patients at increased risk of CVD have difficulty maintaining lifestyle changes and adhering to their medication regimen - either intentionally or unintentionally. Intentional non-adherence could occur when patients experience side-effects of the medication, whereas unintentional non-adherence usually occurs when patients forget to take their medication.

In the current study, the investigators will investigate whether promoting an active choice regarding coping with an increased CVD risk results in better psychological outcomes (e.g., degree of active choice; commitment toward the chosen option) compared to usual care (i.e. a GP's advice to change one's lifestyle and take medication). By 'active choice' the investigators mean a conscious and autonomous choice in which an individual (a) becomes aware of a discrepancy between the current and desired situation; (b) understands what his/her CVD risk means, and what its causes and consequences are; (c) evaluates the pros and cons of the different options to cope with the risk; and (d) is clear about his/her values regarding the choice. The different options to cope with an increased CVD risk include: changing one's lifestyle; taking medication; doing both; or changing nothing.

The investigators will investigate this in a web-based RCT among adults aged 45-65 years. The intervention group (i.e. active choice group) and control group (i.e. usual care group) will both receive a hypothetical CVD risk. The investigators expect an active choice regarding coping with an increased CVD risk to result in better psychological outcomes compared to a GP's advice. Ultimately, a more active choice is expected to results in greater behavioural persistence regarding the chosen option; i.e. lifestyle change and/or medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45-65 years

Exclusion Criteria:

* Suffering/ having suffered from CVD
* Being on lipid lowering or blood pressure lowering medication
* Suffering from diabetes
* kidney damage or rheumatism
* not being able to walk at least 100 meters
* being in a wheelchair
* pregnancy

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators will investigate effect modification by gender. Therefore, the investigators aim to recruit 412 men and 312 women.
Enrollment: 743 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Active choice | Directly after the intervention
  Self-constructed scale. Measures the degree to which participants make an active choice. The scale contains 11 items that have to be answered on a scale of 1 (totally disagree) to 5 (totally agree). A higher mean score on the scale indicates a better outcome.
Intention strength | Directly after the intervention
  2 self-constructed questionnaire items on a scale of 1 (not strong at all) to 10 (very strong). Measure intention strength to perform the chosen behaviour (i.e., lifestyle change and/or taking medication). A higher score indicates a better outcome.
Commitment | Directly after the intervention
  5 self-constructed questionnaire items on a scale of 1 (not at all) to 10 (very much). Measure commitment to perform the chosen behaviour (i.e., lifestyle change and/or taking medication). A higher mean score indicates a better outcome.

SECONDARY OUTCOMES:
Intention | Directly after the intervention
  Self-constructed questionnaire item. Measures intention regarding coping with CVD and intention regarding lifestyle change. 4 options: (a) Lifestyle change; (b) Taking medication; (c) Lifestyle change and taking medication; (d) change nothing.
Self-efficacy | Directly after the intervention
  2 self-constructed questionnaire items on a scale of 1 (not strong at all) to 10 (very strong). Measure self-efficacy regarding performing the chosen option (i.e., lifestyle change and/or taking medication). A higher score indicates a better outcome.
Response efficacy | Directly after the intervention
  2 self-constructed questionnaire items on a scale of 1 (not at all) to 10 (totally). Measure response efficacy regarding coping with an increased CVD risk. A higher mean score indicates a better outcome.
Autonomous motivation subscale of the Treatment Motivation Questionnaire | Directly after the intervention
  6 questionnaire items adapted from the Treatment Motivation Questionnaire (TSRQ). The items measure the degree of autonomous motivation on a scale of 1 (totally disagree) to 7 (totally agree). A higher mean score on this subscale indicates a better outcome.
Knowledge | Directly after the intervention
  4 self-constructed questionnaire items measuring knowledge about CVD. Response options: Agree; Disagree; Don't know.
Cognitive risk perception | Directly after the intervention
  Self-constructed questionnaire item measuring participants' cognitive risk perception. The item has a 5-point scale ranging from 'very small' to 'very big'.
Affective risk perception | Directly after the intervention
  3 self-constructed questionnaire items measuring participants' affective risk perception on a scale of 1 (not at all) to 10 (very much). A higher score indicates more negative emotion associated with the hypothetical risk.
Lifestyle change intention | Directly after the intervention
  Self-constructed questionnaire item. Measures participants' intention regarding lifestyle change. 4 options: Quit smoking; Eat healthier; Become more physically active; Other.

OTHER OUTCOMES:
Perceived Health according to the Research and Development 36 | Directly after the intervention
  Questionnaire item that measures participants' perceived health on a 5-point scale. This is the first item from the questionnaire 'Research and Development 36' (RAND-36). A higher score indicates better perceived health.
Control Preference Scale | Directly after the intervention
  The questionnaire item was adapted from the Control Preferences Scale. A lower score indicates that someone prefers to take decisions himself, whereas a higher score indicates that someone prefers to leave the decision to his doctor.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Timmermans, Prof, Study Director — VU Medical Center, Amsterdam UMC
Locations (1):
- VUMedicalCenter, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be made available online on clinicaltrials.gov. Patient data will only be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol will be permanently available. Participant data will be deleted 15 years after study completion.
Access Criteria: No access restrictions for the study protocol.

REFERENCES:
- [Derived] Landais LL, Jelsma JGM, Damman OC, Verhagen EALM, Timmermans DRM. Fostering active choice to empower behavioral change to reduce cardiovascular risk: A web-based randomized controlled trial. PLoS One. 2024 Aug 1;19(8):e0304897. doi: 10.1371/journal.pone.0304897. eCollection 2024. PMID 39088470

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT05142280/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT05142280/SAP_001.pdf